CLINICAL TRIAL: NCT00120536
Title: Efficacy and Safety of Three Doses of Vildagliptin in Drug Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2384
Record Dates: First submitted 2005-07-12; First posted 2005-07-18 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
The purpose of this study is to assess the long term safety and effectiveness of three doses of vildagliptin, an unapproved drug, compared to placebo in lowering overall blood glucose levels in people with type 2 diabetes who have not previously been treated with drug therapy to lower their blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Not currently on drug therapy for type 2 diabetes
* Blood glucose criteria must be met
* Body mass index (BMI) in the range 22-45

Exclusion Criteria:

* History of type 1 diabetes
* Evidence of significant diabetic complications
* Serious cardiovascular events within the past 6 months
* Laboratory value abnormalities as defined by the protocol
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2005-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 24 weeks

SECONDARY OUTCOMES:
Adverse event profile after 24 weeks of treatment
Change from baseline in fasting plasma glucose at 24 weeks
Patients with endpoint HbA1c < 7% after 24 weeks
Patients with reduction in HbA1c >/= 0.7% after 24 weeks
Change from baseline in HbA1c at 24 weeks for patients with high baseline HbA1c vs. low baseline HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Pratley RE, Schweizer A, Rosenstock J, Foley JE, Banerji MA, Pi-Sunyer FX, Mills D, Dejager S. Robust improvements in fasting and prandial measures of beta-cell function with vildagliptin in drug-naive patients: analysis of pooled vildagliptin monotherapy database. Diabetes Obes Metab. 2008 Sep;10(10):931-8. doi: 10.1111/j.1463-1326.2007.00835.x. Epub 2007 Dec 17. PMID 18093207
- [Derived] Pratley RE, Rosenstock J, Pi-Sunyer FX, Banerji MA, Schweizer A, Couturier A, Dejager S. Management of type 2 diabetes in treatment-naive elderly patients: benefits and risks of vildagliptin monotherapy. Diabetes Care. 2007 Dec;30(12):3017-22. doi: 10.2337/dc07-1188. Epub 2007 Sep 18. PMID 17878242
- [Derived] Pi-Sunyer FX, Schweizer A, Mills D, Dejager S. Efficacy and tolerability of vildagliptin monotherapy in drug-naive patients with type 2 diabetes. Diabetes Res Clin Pract. 2007 Apr;76(1):132-8. doi: 10.1016/j.diabres.2006.12.009. Epub 2007 Jan 12. PMID 17223217